CLINICAL TRIAL: NCT02789150
Title: Outcomes of Renal Function in Hepatorenal Syndrome (HRS) Determined By Comparison of Target Mean Arterial Pressure (MAP) of 65 - 70 Mmhg Versus ≥ 85 Mmhg
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Mohamed Saad, Associate professor of medicine, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14.1190
Record Dates: First submitted 2015-01-28; First posted 2016-06-02 (Estimated); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Hepatorenal Syndrome
MeSH Terms: conditions — Hepatorenal Syndrome | interventions — Norepinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MAP 65-70 (Experimental): Goal MAP of 65-70
  Interventions: Drug: Norepinephrine (Levophed)
- MAP greater than or equal to 85 (Active Comparator): MAP greater than or equal to 85
  Interventions: Drug: Norepinephrine (Levophed)

INTERVENTIONS:
Drug: Norepinephrine (Levophed) — Titrate norepinephrine to MAP 65-70
  Arms: MAP 65-70
Drug: Norepinephrine (Levophed) — Titrate norepinephrine to MAP 85 or greater
  Arms: MAP greater than or equal to 85

SUMMARY:
Comparing renal outcomes based on a Mean Arterail Pressure (MAP) of 65-7085mmhg versus a MAP of greater than or equal to 85mmhg

DETAILED DESCRIPTION:
Main hypothesis:

The investigators propose that there will be no difference clinical outcomes as evidenced by a significant difference in urine output or change in creatinine between the MAP target ≥ 85mmhg and the MAP target of 65-70 mmhg.

Primary end point:

To determine if High MAP or Low MAP will provide the most optimal renal function. The primary endpoints will be 96h UOP and change in creatinine levels. UOP will be calculated as cc/24 hours. The investigators will compare the change in urinary output of day 1 versus day 4. Creatinine will be measured daily and the change from initiation to completion of the study will be recorded. The mean values of these will be compared.

Secondary end point:

To determine if High MAP or Low MAP will decrease the occurrence of cardiac events (arrhythmias and myocardial infarctions) and vascular events (limb or intestinal ischemia).

Study Design:

This is a prospective, unblinded, randomized, Two-arm treatment, pilot study. Patients will undergo block randomization to receive either a MAP ≥ 85mmhg or a MAP 65-70mmhg.

ELIGIBILITY:
Inclusion Criteria:

* 1. Admission to intensive care unit (ICU) 2. Age >18 years old 3. Able to obtain informed consent obtained from the patient, from the patient's power of attorney, or from the next of kin 4. Must meet all major criteria based on the International Ascites Club definition and diagnostic criteria for Hepatorenal Syndrome:

  1. chronic or acute liver disease with advanced hepatic failure and portal hypertension;
  2. the serum creatinine is greater than 1. 5 mg/dL or 24 hour creatinine clearance of less than 40 ml/min;
  3. absence of shock, ongoing bacterial infection, and current or recent treatment with nephrotoxic drugs;
  4. absence of gastrointestinal fluid losses (repeated vomiting or intense diarrhea) or renal fluid losses;
  5. no sustained improvement in renal function defined as a decrease in serum creatinine to less than 1.5 mg/dL or increase in 24 hour creatinine clearance to 40 ml/min or more following diuretic withdrawal and expansion of plasma volume with 1.5 L of isotonic saline;
  6. proteinuria less than 500 mg/dL;
  7. no ultrasonic evidence of obstructive uropathy or parenchymal renal disease. 5. In addition, patients must meet the definition of HRS type I or HRS type I

  <!-- -->

  1. -HRS I defined by a rapid deterioration in kidney function with the serum creatinine increasing by more than 100% from baseline to greater than 2.5mg/dl within a two week period.
  2. -HRS II defined as: patients with refractory ascites with either a steady but moderate degree of functional renal failure (≥ 1.5mg/dl) or deterioration in kidney function that does not fulfill the criteria for HRS type I

Exclusion Criteria:

* 1. pre-existing continuous renal replacement therapy cannot or those initiated on dialysis during their hospital stay.

  2. artificial liver support therapies 3. ongoing gastrointestinal bleeding 4. active surgical issues 5. pre-existing TIPS or TIPS placed during hospital stay 6. long standing hypertension 7. improvement in renal function after central blood volume expansion contraindications to norepinephrine (active myocardial event, ventricular arrhythmia, obstructive physiology, limb ischemia) 8. Pregnancy 9. Treating physicians refusing to enroll patient

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-01; Primary Completion 2018-01-11 (Actual); Study Completion 2018-01-11 (Actual)

PRIMARY OUTCOMES:
Urine output | 2 years
  To determine if High MAP or Low MAP will provide the most optimal renal function. The primary endpoints will be 96h UOP and change in creatinine levels. UOP will be calculated as cc/24 hours. We will compare the change in urinary output of day 1 versus day 4. Creatinine will be measured daily and the change from initiation to completion of the study will be recorded. The mean values of these will be compared.
serum creatinine | 2 years

SECONDARY OUTCOMES:
Cardiac events | 2 years
  To determine if High MAP or Low MAP will decrease the occurrence of cardiac events (arrhythmias and myocardial infarctions) and vascular events (limb or intestinal ischemia).
ischemic events | 2 years
  To determine if High MAP or Low MAP will decrease the occurrence of cardiac events (arrhythmias and myocardial infarctions) and vascular events (limb or intestinal ischemia).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

REFERENCES:
- [Derived] Varajic B, Cavallazzi R, Mann J, Furmanek S, Guardiola J, Saad M. High versus low mean arterial pressures in hepatorenal syndrome: A randomized controlled pilot trial. J Crit Care. 2019 Aug;52:186-192. doi: 10.1016/j.jcrc.2019.04.006. Epub 2019 Apr 15. PMID 31096099